CLINICAL TRIAL: NCT01922375
Title: A Randomized, Double-blind, Double-dummy, Placebo-controlled, Parallel Design Clinical Trial to Evaluate the Efficacy and Safety of Naftopidil in Male Patients With Lower Urinary Tract Symptoms Associated With Benign Prostatic Hyperplasia
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety of Naftopidil in Male Patients With Lower Urinary Tract Symptoms Associated With Benign Prostatic Hyperplasia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dong-A Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Dong-A ST Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FLV_BPH_IV-1
Record Dates: First submitted 2013-02-11; First posted 2013-08-14 (Estimated); Last update posted 2013-08-14 (Estimated); Status verified 2013-08

CONDITIONS: Lower Urinary Tract Symptoms Associated With Benign Prostatic Hyperplasia
MeSH Terms: interventions — naftopidil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Naftopidil dose 2 (Experimental): PO administration
  Interventions: Drug: Naftopidil
- Placebo (Placebo Comparator): PO administration
- Naftopidil dose 1 (Experimental): PO administration
  Interventions: Drug: Naftopidil

INTERVENTIONS:
Drug: Naftopidil
  Arms: Naftopidil dose 1; Naftopidil dose 2

SUMMARY:
This study is designed to evaluate the efficacy and safety of Naftopidil in Korean male patients with with lower urinary tract symptoms associated with benign prostatic hyperplasia.

The investigators hypothesized that Naftopidil which came onto marcket in Japan would effect in improvement of voiding and storage difficulty.

Design:

Placebo-controlled, Randomized, Double-blind, Double-dummy, Parallel group, Fixed dose design

ELIGIBILITY:
Inclusion Criteria:

* Male patients aged 4 years or more diagnosed with BPH

Exclusion Criteria:

* subjects with uncontrolled blood pressure
* subjects with hepatic or renal dysfunction
* subjects with prostate cancer
* Had treatments for BPH using other alpha receptor antagonists within 2 weeks

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 411 (Actual)
Dates: Start 2011-12; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Efficacy(IPSS score change) | From 0 week(baseline) to 12 week(end of the treatment)

SECONDARY OUTCOMES:
Efficacy(IPSS, Uroflowmetry parameter, LUTS-GAQ) | From 0 week(baseline) to 12 week(end of the treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Sae-Woong Kim, MD.PhD, Principal Investigator — Seoul St. Mary's Hospital; Jae-Seok Hyun, Md, PhD, Principal Investigator — Gyeongsang National University Hospital; Du-Geon Moon, MD, PhD, Principal Investigator — Korea University Guro Hospital; Nam-Cheol Park, MD, PhD, Principal Investigator — Pusan National University Hospital; Sung-Won Lee, MD, PhD, Principal Investigator — Samsung Medical Center; Soo-Woong Kim, Md, PhD, Principal Investigator — Seoul National University Hospital; Tai-Young Ahn, Md, PhD, Principal Investigator — Asan Medical Center; Ki-Hak Moon, Md, PhD, Principal Investigator — Yeongnam University Hospital; Woo-Sik Chung, MD,PhD, Principal Investigator — Ewha Womans University Hospital; Kweon-Sik Min, MD, PhD, Principal Investigator — Inje University; Jong Kwan Park, MD, PhD, Principal Investigator — Chonbuk National University Hospital; Dae Yul Yang Yang, MD, PhD, Principal Investigator — Kangdong Sacred Heart Hospital; Ji- Kan Ryu, MD, PhD, Principal Investigator — Inha University Hospital
Locations (1):
- Chonnam national university hospital, Gwangju, South Korea